CLINICAL TRIAL: NCT00539864
Title: Evaluation of Safety and Reactogenicity of FluBlok, Trivalent Recombinant Influenza Vaccine, and Comparison of the Immunogenicity, Efficacy and Effectiveness of FluBlok to a Licensed Egg-Grown Influenza Vaccine in Adults Aged 50 to 64
Brief Title: Safety and Reactogenicity of FluBlok and Comparison of Immunogenicity, Efficacy and Effectiveness Against TIV
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Protein Sciences Corporation (Industry)
Responsible Party: Manon MJ Cox, Protein Sciences Corporation
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: PSC06
Record Dates: First submitted 2007-10-04; First posted 2007-10-05 (Estimated); Results first posted 2011-07-27 (Estimated); Last update posted 2011-07-27 (Estimated); Status verified 2011-07

CONDITIONS: Influenza
Keywords: Influenza
MeSH Terms: conditions — Influenza, Human | interventions — FluBlok; Influenza Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- FluBlok (Experimental): Recombinant Trivalent Hemagglutinin Influenza Vaccine: 2007-2008 formulation containing 45μg of each hemagglutinin derived from A/Solomon Islands/03/2006 (H1N1), A/Wisconsin/67/2005 (H3N2), and B/Malaysia/2506/2004
  135μg total
  Interventions: Biological: FluBlok Influenza Vaccination
- TIV (Fluzone) (Active Comparator): Licensed Trivalent Influenza Vaccine (TIV): 2007-2008 formulation containing 15μg of each hemagglutinin derived from A/Solomon Islands/03/2006 (H1N1), A/Wisconsin/67/2005 (H3N2), and B/Malaysia/2506/2004
  45μg total
  (Fluzone, sanofi pasteur)
  Interventions: Biological: TIV (Fluzone) Influenza Vaccination

INTERVENTIONS:
Biological: FluBlok Influenza Vaccination — 0.5mL dose for intramuscular injection
  Other Names: FluBlok; rHA; rHA0; recombinant hemagglutinin
  Arms: FluBlok
Biological: TIV (Fluzone) Influenza Vaccination — 0.5mL dose for intramuscular injection
  Other Names: Fluzone; TIV
  Arms: TIV (Fluzone)

SUMMARY:
The purpose of this study was to evaluate and compare the safety, reactogenicity, immunogenicity, relative efficacy and effectiveness of FluBlok to a licensed trivalent influenza vaccine (TIV)in healthy adults age 50-64 years.

DETAILED DESCRIPTION:
Annual influenza epidemics are associated with serious excess morbidity and mortality, particularly among the elderly. Licensed trivalent inactivated influenza vaccines (TIVs) have been shown to reduce hospitalization and death following influenza in this vulnerable population, but their efficacy is lower than that observed in younger, healthy populations. In addition, recent studies have questioned the level of effectiveness of TIV in the elderly, suggesting that cohort studies have overestimated the benefits of immunization with current TIV formulations in this age group. In view of these considerations, it is widely accepted that improved and alternative vaccines are needed for control of seasonal and pandemic influenza.

Currently available TIVs are prepared from viruses that are grown in embryonated hens' eggs. Alternative substrates for vaccine production are desirable in order to reduce the vulnerability of and to expand influenza vaccine supply. Recombinant DNA techniques allow for expression of the influenza hemagglutinin (rHA) by baculovirus vectors in insect cell cultures. Advantages of this technique include speed of production, absence of egg protein, and a highly purified product. Previous studies among healthy younger and older adults have confirmed that rHA vaccines are safe, well tolerated and immunogenic at dosages up to nine times higher than those contained in TIV. Dose-related increases in serum antibody levels after immunization also were observed.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 50 to 64.
* Females should be at least 2 years post-menopausal or sterile or practicing accepted form of birth control (including: condom with spermicidal, licensed hormonal contraceptive, abstinence, IUD or monogamous relationship with a vasectomized partner).
* Healthy, as determined by oral temperature <100.0°F, medical history, and medical assessment w/ brief physical evaluation by RN (if indicated) based on medical history.
* Able to understand and comply with planned study procedures.
* Provides written informed consent prior to initiation of any study procedure.

Exclusion Criteria:

* Known allergy to eggs or other vaccine components.
* Immunosuppression as a result of an underlying illness or treatment, or used anticancer chemotherapy or radiation therapy within the preceding 36 months.
* Any malignancy other than localized prostate cancer, diagnosed or treated actively during the past 5 years. Exceptions: Subjects with a history of lymphoproliferative disorder at any time in their life will be excluded, while subjects with a history of localized nonmelanotic skin cancer that has been completely removed during the past 5 years may be eligible.
* Long-term use of oral steroids, parenteral steroids, or high-dose inhaled steroids (>800 mcg/day of beclomethasone dipropionate or equivalent) within the preceding 6 months (Nasal and topical steroids are allowed).
* Diagnosis of or treatment for bipolar disorder, severe major depression, schizophrenia or other major psychotic disorder in the past 3 months that is associated with severely impaired judgment or cognition.
* History of receiving immunoglobulin or other blood product within the 3 months prior to enrollment in this study.
* Receipt of any other licensed vaccines within 2 weeks (for inactivated vaccines) or 4 weeks (for live vaccines) prior to enrollment in this study.
* Use of experimental vaccines or any influenza vaccine other than FluBlOk after May 31st 2007 for the 2008 Southern Hemisphere or 2007 to 2008 Northern hemisphere epidemic seasons.
* History of severe reactions following immunization with influenza virus vaccines.
* Moderate to severe acute illness or febrile illness (oral temperature greater than 100degreesF) within 1 week prior to vaccination.
* Receipt of an experimental agent (vaccine, drug, biologic, device, blood product or medication) within 1 month prior to enrollment in this study, or expects to receive an experimental agent during study period.
* Known active human immunodeficiency virus, hepatitis B, or hepatitis C infection.
* History of alcohol or drug abuse in the last 5 years.
* History of Guillain-Barré Syndrome.
* Subject is not available for three (3) or more consecutive weeks during active influenza season.
* Any acute or chronic medical condition that, in the opinion of the investigator, would render vaccination unsafe, interfere with the evaluation of responses, or render the subject unable to meet the requirements of the protocol. These conditions include, but are not limited to: history of significant renal impairment (dialysis and treatment for kidney disease, including diabetic and hypertensive kidney disease); subjects with diabetes mellitus, well-controlled with oral agents may enroll as long there has been no dosage increase within the past 6 months; insulin-dependent diabetes is excluded; cardiac insufficiency, if heart failure is present (New York Heart Association Functional Class III or IV); an arteriosclerotic event during the 6 months prior to enrollment (e.g., history of myocardial infarction, stroke, recanalization of femoral arteries, or transient ischemic attack)

Ages: 50 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 602 (Actual)
Dates: Start 2007-09; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roger Baxter, MD, Principal Investigator — Kaiser Permanenter Center for Vaccine Development
Locations (5):
- United States (5):
  - Kaiser Permanente Pediatric Clinic - Fresno, Fresno, California
  - Kaiser Permanente Pediatric Clinic - Hayward, Hayward, California
  - Kaiser Permanente Pediatric Clinic - Roseville, Roseville, California
  - Kaiser Permanente Pediatric Clinic - Sacramento, Sacramento, California
  - Kaiser Permanente, Honolulu, Hawaii

REFERENCES:
- [Result] Baxter R, Patriarca PA, Ensor K, Izikson R, Goldenthal KL, Cox MM. Evaluation of the safety, reactogenicity and immunogenicity of FluBlok(R) trivalent recombinant baculovirus-expressed hemagglutinin influenza vaccine administered intramuscularly to healthy adults 50-64 years of age. Vaccine. 2011 Mar 9;29(12):2272-8. doi: 10.1016/j.vaccine.2011.01.039. Epub 2011 Jan 28. PMID 21277410
- See also: Related Info — http://proteinsciences.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects 50 - <64 years of age were screened in participating outpatient clinics for eligibility within 30 days of randomization during the 2007 influenza season.
Pre-assignment Details: Subjects whose laboratory values were exclusionary were not randomized. Women of child-bearing potential were required to have a negative pregnancy test.
Period: Overall Study
Arm/Group | FluBlok | TIV (Fluzone)
Started | 300 | 302
Completed | 299 | 300
Not Completed | 1 | 2
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | FluBlok | TIV (Fluzone) | Total
Number analyzed (Participants) | 300 | 302 | 602
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 300 | 302 | 602
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 55.9 (3.71) | 55.7 (3.64) | 55.8 (3.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 187 | 192 | 379
  Male | 113 | 110 | 223
Region of Enrollment [Number; unit: participants]
  United States | 300 | 302 | 602

OUTCOME MEASURES:

1. Secondary Outcome: Evaluation and Comparison of Immunogenicity of FluBlok and TIV in Healthy Adults 50-64 Years of Age.
Description: Immunogenicity was assessed by measuring the difference in values in Hemagglutination-Inhibition Assay (HAI) titers in participants from Day 0 to Day 28, using Geometric Mean Titers (GMTs). The GMTs from the FluBlok and TIV groups were then compared.
Time Frame: Day 0 and Day 28
Population: All randomized subjects who received study vaccine and had Day 0 and Day 28 HAI titers
Measure: Geometric Mean (95% Confidence Interval); unit: HAI Titers
Arm/Group | FluBlok | TIV (Fluzone)
Number analyzed (Participants) | 299 | 302
HAI Titers
  A/Solomon Islands (H1N1) - Day 0 | 28.71 [25.59 to 32.21] | 27.77 [25.07 to 30.76]
  A/Solomon Islands (H1N1) - Day 28 | 181.34 [159.61 to 206.02] | 139.74 [124.64 to 156.66]
  A/Wisconsin (H3N2) - Day 0 | 18.57 [16.37 to 21.06] | 18.20 [16.07 to 20.62]
  A/Wisconsin (H3N2) - Day 28 | 105.41 [91.01 to 122.09] | 60.88 [53.58 to 69.18]
  B/Malaysia - Day 0 | 48.49 [43.38 to 54.19] | 49.18 [43.77 to 55.25]
  B/Malaysia - Day 28 | 110.93 [100.07 to 122.97] | 116.03 [104.16 to 129.25]

2. Primary Outcome: Number of Participants With Reactogenicity (Solicited) Adverse Events (AEs)
Description: Solicited reactogenicity events included injection site pain, bruising, erythema and swelling. Solicited systemic AEs included fatigue, chills, arthralgias, myalgias, headache and nausea.
Time Frame: Reactogenicity days 0-7 following immunization; other AEs days 0-28 following immunization
Population: Safety population included all randomized subjects who received a dose of study vaccine.
Measure: Number; unit: participants
Arm/Group | FluBlok | TIV (Fluzone)
Number analyzed (Participants) | 300 | 302
participants
  Fatigue | 40 | 62
  Chills | 12 | 15
  Arthralgias | 15 | 19
  Myalgia | 40 | 63
  Headache | 59 | 63
  Nausea | 13 | 15
  Injection Site Pain | 154 | 165
  Injection Site Bruising | 16 | 14
  Injection Site Erythema | 24 | 25
  Injection Site Swelling | 25 | 30

3. Secondary Outcome: Percentage of Participants With Seroconversion
Description: Percentage of participants with greater than or equal to a 4-fold rise in Hemagglutination-Inhibition Assay (HAI) titer over Day 0 at Day 28 following immunization
Time Frame: Day 28 following immunization at Day 0
Population: All randomized subjects who received study vaccine and who had day 0 and day 28 HAI titers
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Units Other Than Participants: % of participants
Arm/Group | FluBlok | TIV (Fluzone)
Number analyzed (Participants) | 299 | 302
Number analyzed (% of participants) | 100 | 100
Percentage of participants
  A/Solomon Islands (H1N1) | 72 [66.8 to 77.2] | 66 [60.6 to 71.5]
  A/Wisconsin (H3N2) | 61 [55.4 to 66.8] | 44 [38.0 to 69.2]
  B/Malaysia | 41 [35.2 to 46.6] | 41 [35.5 to 46.8]

4. Secondary Outcome: Percentage of Participants With Seroprotection
Description: Percentage of participants with (HAI titer greater than or equal to 40) at Day 28
Time Frame: Day 28 following immunization at Day 0
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | FluBlok | TIV (Fluzone)
Number analyzed (Participants) | 300 | 302
Percentage of participants
  Influenza A/Solomon Islands (H1N1) | 96 [93.5 to 98.1] | 96 [92.8 to 97.7]
  Influenza A/Wisconsin (H3N2) | 85 [80.8 to 89.1] | 75 [69.9 to 79.9]
  Influenza B/Malaysia | 93 [89.5 to 95.6] | 94 [91.1 to 96.7]

ADVERSE EVENTS:
Time Frame: All AEs - 28 days following immunization; SAEs for duration of influenza season.
Arm/Group | FluBlok | TIV (Fluzone)
Serious Adverse Events (participants affected / at risk) | 1/300 | 0/302
Other Adverse Events (participants affected / at risk) | 4/300 | 9/302
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FluBlok (N=300) | TIV (Fluzone) (N=302)
Vasovagal Syncope (Cardiac disorders) | 1 (1) | 0 (0) — Subject experienced a syncopal episode, was treated with intravenous fluids in ER and discharged home without sequelae.
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FluBlok (N=300) | TIV (Fluzone) (N=302)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 9 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No